CLINICAL TRIAL: NCT02515032
Title: A 12-week Double Blind, Placebo Controlled, Randomised Pilot Study Assessing Safety and Tolerability of Nutrifriend Cachexia in Patients Diagnosed With Non Small Cell Lung Cancer (NSCLC) With Involuntary Weight Loss
Brief Title: Pilot Study of Safety and Tolerability of Nutrifriend Cachexia in NSCLC Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smartfish AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF-C002
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Cachexia; NSCLC
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NF Cachexia (Experimental): Nutrifriend Cachexia, an Omega-3 enriched fruit juice (non complete dietary formula).
  Interventions: Dietary Supplement: Nutrifriend Cachexia
- Placebo (Placebo Comparator): An isocaloric placebo comparator
  Interventions: Dietary Supplement: Isocaloric placebo

INTERVENTIONS:
Dietary Supplement: Nutrifriend Cachexia — 2 daily for 12 weeks
  Other Names: NFCax
  Arms: NF Cachexia
Dietary Supplement: Isocaloric placebo — 2 daily for 12 weeks
  Other Names: Placobo
  Arms: Placebo

SUMMARY:
SF-C002 is a pilot study in patients with newly diagnosed NSCLC suffering from involuntary weight loss. The study is 12 weeks, double-blinded, placebo controlled and the main objective is to study the safety and tolerability of Nutrifriend Cachexia.

DETAILED DESCRIPTION:
This study is a 12-week, randomised, parallel group, placebo controlled, multi-centre study. The primary objective is to evaluate the safety and tolerability of Nutrifriend Cachexia in patients with NSCLC. The secondary objectives of the study are to evaluate effects on body composition, muscle function, daily activity, inflammation, tumor growth, compliance, appetite and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* First-line standard chemotherapy as curative or palliative treatment for NSCLC
* Will start the first cycle of standard chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Involuntary weight loss

Exclusion Criteria:

* Another invasive malignancy in the last 2 years.
* Previous relapse of NSCLC within 2 years of randomisation
* Other cachectic disorders such as renal or hepatic disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by (adverse events, concomitant medication and laboratory markers) of Nutrifriend Cachexia in patients with NSCLC | 12 weeks

SECONDARY OUTCOMES:
Body composition assessed by fat mass and lean body mass (LBM) | 12 weeks
Body composition assessed by weight | 12 weeks
Body composition assessed by BMI | 12 weeks
Body composition assessed by waist circumference | 12 weeks
Body composition assessed by calf circumference | 12 weeks
Function assessed by 6 minute walking test | 12 weeks
Function assessed by grip strength | 12 weeks
Function assessed by walking distance | 12 weeks
Inflammation | 12 weeks
  IL-6, IL-8, TNF-alpha, CRP
Metabolic markers | 12 weeks
  Glucose, insulin, cholesterol, HbA1c
QoL assessed by EORTC QLQ-C3 | 12 weeks
QoL assessed by Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire | 12 weeks
QoL assessed by Nutrition Appetite Questionnaire (CNAQ) | 12 weeks
Compliance assessed by Drinks consumed | 12 weeks
Compliance assessed by vitamin D levels | 12 weeks
Compliance assessed by Omega-3 incorporation | 12 weeks

OTHER OUTCOMES:
Response to chemotherapy by tumor growth | 12 weeks
Overall survival | 52 weeks
Exploratory biomarkers related to cachexia, e.g. carnosine, beta-alanine | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Muscaritoli, Prof., Principal Investigator — University Hospital Sapienza
Locations (14):
- Croatia (4):
  - GH Varaždin, Varaždin
  - GH Zadar, Zadar
  - CHC Sestre Milosrdnice, Zagreb
  - CHC Zagreb,, Zagreb
- Italy (3):
  - Policlinico Universitario Campus Bio-Medico di Roma, Rome
  - Policlinico Tor Vergata, Rome
  - Azienda Ospedaliera San Camillo Forlanini, Rome
- Slovakia (5):
  - FNsP F.D. Roosvelta Banská Bystrica, Banská Bystrica
  - Nemocnica Sv. Jakuba, Bardejov
  - Východoslovenský onkologický ústav, Košice
  - NsP Štefana Kukuru Michalovce, Michalovce
  - FNsP J.A. Reimana, Prešov
- Sweden (2):
  - Linkoping University Hospital, Linköping
  - Akademiska hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laviano A, Calder PC, Schols AMWJ, Lonnqvist F, Bech M, Muscaritoli M. Safety and Tolerability of Targeted Medical Nutrition for Cachexia in Non-Small-Cell Lung Cancer: A Randomized, Double-Blind, Controlled Pilot Trial. Nutr Cancer. 2020;72(3):439-450. doi: 10.1080/01635581.2019.1634746. Epub 2019 Jul 10. PMID 31290697